CLINICAL TRIAL: NCT01701063
Title: A Two-Part, Open-Label, Single-Arm Phase 1/2 Study of Safety, Pharmacokinetics, and Efficacy of Telaprevir in Combination With Peginterferon Alfa-2b and Ribavirin in Pediatric Subjects Aged 3 to 17 Infected With Genotype 1 Hepatitis C Virus
Brief Title: An Open-Label Study of the Effect of Telaprevir in Combination With Peginterferon Alfa-2b and Ribavirin in Pediatric Subjects Infected With Hepatitis C Virus
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX11-950-118
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment-Naive or Prior Partial/Null Response (Experimental): telaprevir + Peginterferon alfa-2b + Ribavirin
  Interventions: Drug: Telaprevir; Drug: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — 100- and 250-mg chewable tablets or 375-mg film-coated tablets for oral administration
Drug: Peginterferon alfa-2b — 50 μg/0.5 mL, 80 μg/0.5 mL, 120 μg/0.5 mL, or 150 μg/0.5 mL for subcutaneous (SC) injection
  Other Names: PegIntron®
Drug: Ribavirin — 200-mg capsules or 40-mg/mL solution for oral administration
  Other Names: Rebetol®

SUMMARY:
The purpose of this study is to assess the safety, efficacy, and pharmacokinetics in a carefully monitored cohort of pediatric subjects infected with hepatitis C virus (HCV) on a telaprevir-based regimen in Part A and with dose adjustments if needed before Part B.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 3 to 17 years of age
* Chronic hepatitis C
* Hepatitis C virus genotype 1a or b at the Screening Visit
* Subject is judged to be in good health (besides HCV infection) in the opinion of the investigator.
* Signed informed consent form (ICF), and where appropriate, signed Assent Form

Exclusion Criteria:

* History of or prior evidence of a medical condition associated with chronic liver disease other than HCV
* Body weight <15 kg or >90 kg
* Prior evidence of hepatic decompensation
* Contraindications to pegylated interferon/ribavirin (Peg-IFN/RBV)
* History or other evidence of severe retinopathy or clinically significant ophthalmological disorder
* History of non-genotype 1 HCV
* Participation in investigational drug study as described in Study Protocol
* Use of prohibited drugs within 7 days or 5 half-lives before the first dose of study drug

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (23):
- United States (13):
  - Phoenix, Arizona
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - New York, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Seattle, Washington
- Brussels, Belgium
- Wuppertal, Germany
- Italy (3):
  - Milan
  - Padua
  - Pisa
- Spain (2):
  - Esplugues de Llobregat
  - Madrid
- United Kingdom (3):
  - Birmingham
  - Leeds
  - London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 parts (Part A and Part B), which would use separate groups of participants. However, the study was terminated early (12 weeks after last dose of study drug in Part A) and Part B was not conducted.
Groups:
- Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV: Participants aged 13 to 17 years received telaprevir twice daily for 12 weeks either as a film coated tablet (15 milligram per kilogram [mg/kg] of body weight) or as a chewable tablet (14 mg/kg of body weight) in combination with pegylated interferon alfa 2b (Peg-IFN-alfa-2b) 60 microgram per meter square (mcg/m^2) subcutaneous injection weekly and ribavirin (RBV) 200 mg capsules or 40 milligram per milliliter (mg/mL) solution orally twice daily with a maximum dose of 1200 mg per day. Peg-IFN-alfa-2b and RBV were administered for 24 weeks in participants who achieved extended rapid virologic response (eRVR) or for 48 weeks in participants who did not achieve eRVR. eRVR was defined as undetectable hepatitis C virus ribonucleic acid (HCV RNA) levels at Week 4 and Week 12.
- Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV: Participants aged 7 to 12 years received telaprevir twice daily for 12 weeks as a chewable tablet (16 mg/kg of body weight) in combination with Peg-IFN-alfa-2b 60 mcg/m^2 subcutaneous injection weekly and RBV 200-mg capsules or 40 mg/mL solution orally twice daily with a maximum dose of 1200 mg per day. Peg-IFN-alfa-2b and RBV were administered for 24 weeks in participants who achieved eRVR or for 48 weeks in participants who did not achieve eRVR. eRVR was defined as undetectable HCV RNA levels at Week 4 and Week 12.
- Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV: Participants aged 3 to 6 years received telaprevir twice daily for 12 weeks as a chewable tablet (18 mg/kg of body weight) in combination with Peg-IFN-alfa-2b 60 mcg/m^2 subcutaneous injection weekly and RBV 200-mg capsules or 40 mg/mL solution orally twice daily with a maximum dose of 1200 mg per day. Peg-IFN-alfa-2b and RBV were administered for 24 weeks in participants who achieved eRVR or for 48 weeks in participants who did not achieve eRVR. eRVR was defined as undetectable HCV RNA levels at Week 4 and Week 12.
Period: Overall Study
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Started | 13 | 19 | 10
Completed | 13 | 18 | 8
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV: Participants aged 13 to 17 years received telaprevir twice daily for 12 weeks either as a film coated tablet (15 mg/kg of body weight) or as a chewable tablet (14 mg/kg of body weight) in combination with Peg-IFN-alfa-2b 60 mcg/m^2 subcutaneous injection weekly and RBV 200 mg capsules or 40 mg/mL solution orally twice daily with a maximum dose of 1200 mg per day. Peg-IFN-alfa-2b and RBV were administered for 24 weeks in participants who achieved eRVR or for 48 weeks in participants who did not achieve eRVR. eRVR was defined as undetectable HCV RNA levels at Week 4 and Week 12.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Total
Number analyzed (Participants) | 13 | 19 | 10 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (2.06) | 10.2 (1.57) | 4.9 (0.88) | 10.4 (4.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 4 | 28
  Male | 2 | 6 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from the participant's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents administered during the course of the study.
Time Frame: Baseline up to Week 52
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 19 | 10
participants
  Participants with SAEs | 0 | 0 | 1
  Participants with AEs | 13 | 18 | 10

2. Secondary Outcome: Percentage of Participants With Sustained Viral Response 12 Weeks After Last Planned Dose of Study Drug (SVR12)
Description: SVR12 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (less than [<] lower limit of quantification) at 12 weeks after last planned dose of study drug. The plasma HCV RNA level was measured using Roche COBAS TaqMan HCV/High Pure System (HPS) RNA assay version 2.0. The lower limit of quantification was 25 international units per milliliter (IU/mL).
Time Frame: 12 weeks after last planned dose of study drug (up to Week 60)
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 19 | 10
percentage of participants | 69.2 | 89.5 | 40.0

3. Secondary Outcome: Percentage of Participants With Sustained Viral Response 24 Weeks After Last Planned Dose of Study Drug (SVR24)
Description: SVR24 was defined as an undetectable HCV RNA Levels (< lower limit of quantification) at 24 weeks after last planned dose of study drug. The plasma HCV RNA level was measured using Roche COBAS TaqMan HCV/HPS RNA assay version 2.0. The lower limit of quantification was 25 IU/mL.
Time Frame: 24 weeks after last planned dose of study drug (up to Week 72)
Population: SVR24 was not analyzed because study was terminated early and follow-up was conducted only up to 12 weeks after planned end of treatment (EOT).
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: The plasma HCV RNA level was measured using Roche COBAS TaqMan HCV/HPS RNA assay version 2.0. The lower limit of quantification was 25 IU/mL. RVR was defined as an undetectable HCV RNA (<lower limit of quantification) 4 weeks after the start of study treatment.
Time Frame: Week 4
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 19 | 10
percentage of participants | 69.2 | 73.7 | 70.0

5. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: The plasma HCV RNA level was measured using Roche COBAS TaqMan HCV/HPS RNA assay version 2.0. The lower limit of quantification was 25 IU/mL. eRVR was defined as an undetectable HCV RNA (<lower limit of quantification) at both 4 weeks and 12 weeks after the start of study treatment.
Time Frame: Week 4 and Week 12
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 19 | 10
percentage of participants | 61.5 | 73.7 | 60.0

6. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA at Week 12
Description: The plasma HCV RNA level was measured using Roche COBAS TaqMan HCV/HPS RNA assay version 2.0. The lower limit of quantification was 25 IU/mL.
Time Frame: Week 12
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 19 | 10
percentage of participants | 69.2 | 89.5 | 70.0

7. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On treatment virologic failure was defined as meeting any futility rule or completing assigned treatment duration and having detectable HCV RNA at EOT. The plasma HCV RNA level was measured using Roche COBAS TaqMan HCV/HPS RNA assay Version 2.0. The lower limit of quantification was 25 IU/mL. Futility rules: 1) HCV RNA >1000 IU/mL at Week 4; 2) HCV RNA >1000 IU/mL at Week 12; 3) Detectable HCV RNA after Week 12 to end of treatment.
Time Frame: Baseline up to Week 48
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 19 | 10
percentage of participants | 15.4 | 5.3 | 30.0

8. Secondary Outcome: Percentage of Participants With Virologic Relapse
Description: The plasma HCV RNA level was measured using Roche COBAS TaqMan HCV/HPS RNA assay Version 2.0. The lower limit of quantification was 25 IU/mL. Viral relapse was defined as having detectable HCV at follow-up in participants who had HCV RNA less than (<) lower limit of quantification (LLOQ) at planned EOT.
Time Frame: 12 weeks after planned EOT (up to Week 60)
Population: FAS included all enrolled participants who received at least 1 dose of study drug. Here 'Number of Participants Analyzed' signifies those participants who completed the assigned treatment period and had undetectable HCV RNA at EOT.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 9 | 17 | 7
percentage of participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Telaprevir Resistant HCV Variant at Non-Structural Viral Protein 3-4A (NS3-4A) Region
Description: Sequence analysis of the HCV NS3-4A region was performed to monitor telaprevir-resistant variants. HCV RNA was isolated from the plasma, amplified by reverse transcription-polymerase chain reaction (RT-PCR), and sequenced (sequencing assay limit of detection HCV RNA >=1000 IU/mL). Results of this outcome measure were to be reported for overall participants instead of by age.
Time Frame: Baseline, On treatment (up to Week 48)
Population: FAS. Here 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome and 'n' signifies those who were evaluable at the specified time point.
Measure: Number; unit: participants
Groups:
- Overall Participants: Participants aged 3 to 17 years received telaprevir twice daily for 12 weeks either as a film coated tablet (15 mg/kg of body weight) or as a chewable tablet (14 to 18 mg/kg of body weight) in combination with Peg-IFN-alfa-2b 60 mcg/m^2 subcutaneous injection weekly and RBV 200 mg capsules or 40 mg/mL solution orally twice daily with a maximum dose of 1200 mg per day. Peg-IFN-alfa-2b and RBV were administered for 24 weeks in participants who achieved eRVR or for 48 weeks in participants who did not achieve eRVR. eRVR was defined as undetectable HCV RNA levels at Week 4 and Week 12.
Arm/Group | Overall Participants
Number analyzed (Participants) | 41
participants
  Baseline (n = 41) | 2
  On treatment (n = 6) | 6

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Telaprevir
Description: Cmax was measured for telaprevir only.
Time Frame: Cohort 1: Pre-dose and 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, and 8.0 hours post-dose on Day 7, Cohort 2: Pre-dose and 0.5, 2.0, 4.0, 5.0, 6.0, and 8.0 hours post-dose on Day 7, Cohort 3: Pre-dose and 1.5, 4.0, and 8.0 hours post-dose on Day 7
Population: Pharmacokinetic (PK) population included all participants who received at least a single dose of telaprevir, whether the participant completed all treatments or not. Here 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 13 | 9
nanogram per milliliter (ng/mL) | 4310 (1160) | 5050 (884) | 4060 (1500)

11. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Telaprevir
Description: Tmax was measured for telaprevir only.
Time Frame: as for outcome 10
Population: PK population. Here 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 13 | 9
hours (h) | 4.00 [1.92 to 8.00] | 4.00 [1.98 to 6.02] | 4.00 [1.50 to 8.00]

12. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Telaprevir
Description: AUC was measured for telaprevir only. AUC 0-t last was defined as the area under the concentration-time curve from the time of dosing to the last measurable concentration. AUC 0-12 hour (AUC 0-12h) was calculated by respecifying predose concentrations as 12 hour concentrations. AUC 0-24h was calculated as AUC 0-12h multiplied by 2. Dose adjusted AUC (AUC 0-24h_Adj) was calculated by multiplying AUC 0-24h by the dose adjustment factor to obtain projected exposures in participants who were misdosed. Data were presented for AUC 0-t last, AUC 0-12h, AUC 0-24h, AUC 0-24h_Adj.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 13 | 13 | 9
hours*nanogram per milliliter (h*ng/mL)
  AUC 0-t last | 39900 (11300) | 43300 (9480) | 35300 (12000)
  AUC 0-12h | 39900 (11300) | 44100 (9020) | 35300 (12000)
  AUC 0-24h | 79900 (22700) | 88100 (18000) | 70600 (24100)
  AUC 0-24h_Adj | 95700 (29800) | 88600 (19200) | 76300 (22800)

13. Secondary Outcome: Elimination Half-Life (T1/2) of Telaprevir
Description: T1/2 was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: as for outcome 10
Population: Half life was not calculated because the calculation required the slope of terminal elimination phase and the PK sampling was relatively sparse and did not yield a terminal elimination phase from which half-life can be accurately estimated.
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Arm/Group | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/19 | 1/10
Other Adverse Events (participants affected / at risk) | 13/13 | 18/19 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV (N=13) | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV (N=19) | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV (N=10)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (13-17 Years): Telaprevir + Peg-IFN-alfa-2b + RBV (N=13) | Cohort 2 (7-12 Years): Telaprevir + Peg-IFN-alfa-2b + RBV (N=19) | Cohort 3 (3-6 Years): Telaprevir + Peg-IFN-alfa-2b + RBV (N=10)
Vomiting (Gastrointestinal disorders) | 8 (13) | 12 (23) | 6 (12)
Nausea (Gastrointestinal disorders) | 7 (9) | 5 (9) | 5 (14)
Anal pruritus (Gastrointestinal disorders) | 4 (6) | 4 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (9) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (6) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (35) | 11 (38) | 8 (75)
Fatigue (General disorders) | 7 (7) | 5 (11) | 3 (7)
Pain (General disorders) | 2 (6) | 4 (8) | 5 (23)
Injection site erythema (General disorders) | 3 (3) | 2 (2) | 3 (5)
Influenza like illness (General disorders) | 1 (1) | 2 (3) | 1 (2)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (2)
Discomfort (General disorders) | 1 (2) | 2 (10) | 0 (0)
Injection site pruritus (General disorders) | 1 (2) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (4) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (3) | 0 (0) | 0 (0)
Product taste abnormal (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (31) | 16 (79) | 6 (12)
Dizziness (Nervous system disorders) | 5 (7) | 5 (6) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (10) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (8) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parvovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 5 (5) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (5) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 5 (6) | 3 (3)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Mood altered (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Flat affect (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep terror (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (6) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 2 (6)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (3) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early because it was determined that telaprevir/Peg-IFN/RBV regimen did not present a meaningful therapeutic treatment over existing interferon-free regimens and was unlikely to be used for participants aged 3 to 17 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.